CLINICAL TRIAL: NCT05683418
Title: A Study to Evaluate the Safety and Tolerability of the Covalent Phosphoinositide-3-Kinase (PI3K)-Alpha Inhibitor, TOS-358, in Adult Subjects With Select Solid Tumors
Brief Title: A Study to Evaluate the Safety and Tolerability of TOS-358 in Adults With HR+ Breast Cancer and Other Select Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Totus Medicines (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOS-358-001; 2023-505346-26-01 (EU CTIS Number)
Record Dates: First submitted 2022-11-12; First posted 2023-01-13 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Squamous Cell Carcinoma of Head and Neck; Endometrial Cancer; HR+/HER2-negative Breast Cancer; Bladder Cancer
Keywords: PI3K-alpha
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Endometrial Neoplasms; Urinary Bladder Neoplasms; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Intervention Model Description: TOS-358 Single Agent Arm:
  Part 1 (multiple ascending doses, QD or BID): locally advanced, recurrent or metastatic HR+ breast, endometrial, urothelial or squamous cell carcinoma of the head and neck, with PIK3CA mutation per local assessment; Part 2 (RP2D determined in Part 1) Patients with locally advanced, recurrent or metastatic HR+ breast cancer with PIK3CA mutation per local assessment will be enrolled protocol defined groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TOS-358 Single Agent Arm (Experimental): Multiple doses of TOS-358 for oral administration.
  Interventions: Drug: TOS-358

INTERVENTIONS:
Drug: TOS-358 — Covalent Phosphoinositide-3-Kinase (PI3K)-alpha Inhibitor

SUMMARY:
The goal of this clinical trial is to evaluate the safety of TOS-358 in adults with select solid tumors who meet study enrollment criteria. The main questions it aims to answer are:

1. what is the maximum tolerated dose and recommended dose for phase 2?
2. how safe and tolerable is TOS-358 at different dose levels when taken orally once or twice per day?

DETAILED DESCRIPTION:
This study will be conducted in two parts: a dose finding portion to determine the maximum tolerated dose and recommended phase 2 dose (RP2D) of TOS-358 administered orally on once a day (QD) and twice daily (BID) schedules, and a dose expansion portion to evaluate safety and tolerability in tumor-specific cohorts administered TOS-358 at the recommended phase 2 dose and schedule.

Adult subjects with histologically confirmed diagnosis of hormone receptor-positive (HR+), human epidermal growth factor receptor 2 (HER2) negative breast cancer, squamous cell carcinoma of the head and neck, cancer of the bladder, or endometrial cancer with known PIK3CA mutations or amplifications and who meet all of the eligibility criteria will be enrolled in the study.

In the dose finding portion of the study, TOS-358 will be evaluated as a single-agent at multiple dose levels administered orally until disease progression, unacceptable toxicity, or until meeting any other reason for discontinuation as specified in the protocol.

ELIGIBILITY:
Key Inclusion Criteria

* Locally advanced, recurrent, or metastatic, incurable (any number of previous lines of therapy is allowed), histologically or cytologically confirmed; HR +/HER2- breast cancer; squamous cell carcinoma of the head and neck; urothelial cancer; or endometrial cancer with no more than 3 prior lines of therapy for metastatic disease
* Willing and able to provide written informed consent for this study
* Adults ≥ 18 years old at time of consent
* Known PIK3CA mutations or amplifications as determined at a CAP/CLIA-certified or equivalently accredited diagnostic laboratory using a validated test
* Measurable disease by RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy ≥ 6 months, as determined by the investigator
* Adequate bone marrow, liver, and kidney function within 14 days prior to first dose of investigational product
* Fasting plasma glucose <= 140 mg/dL AND hemoglobin A1c (HbA1c) <= 7.0%
* Available archived or fresh tumor tissue sample for detection of PIK3CA mutation by central laboratory test

Key Exclusion Criteria

* Recent systemic anticancer treatment prior to start of treatment (EXCEPTION: Patients with breast cancer who were receiving a fulvestrant-containing regimen at the time of informed consent may remain on fulvestrant while receiving study treatment)
* For non-breast cancer: prior treatment with any PI3K, AKT, or mTOR inhibitor, or any agent whose mechanism of action is to inhibit the PI3K-AKT-mTOR pathway,
* Has an established diagnosis of diabetes mellitus type 1 or has uncontrolled diabetes mellitus type 2 requiring antihyperglycemic medication
* Known active central nervous system (CNS) metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Determine the rate of dose-limiting toxicities (DLTs) | First 21 days of treatment
Incidence and severity of adverse events (AEs) and specific laboratory abnormalities graded according to NCI CTCAE v5 | Start of treatment to 30 days after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Zelanna Goldberg, MD, Study Director — Totus Medicines
Locations (18):
- United States (9):
  - University of Southern California, Norris Comprehensive Cancer Center, Los Angeles, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
- Spain (9):
  - NEXT Oncology - Hospital Quironsalud Barcelona - PPDS, Barcelona
  - START Barcelona HM Nou Delfos, Barcelona
  - Instituto de Investigacion Oncologica Vall dHebron (VHIO) - EPON, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - START MADRID Hospital Universitario Fundacion Jimenez Diaz - EDOS, Madrid
  - START MADRID Hospital Universitario HM Sanchinarro - CIOCC, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - NEXT Oncology - Hospital Quironsalud Madrid - PPDS, Pozuelo de Alarcón
  - Hospital Clinico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No